CLINICAL TRIAL: NCT05144243
Title: A Phase 4 Study of Venetoclax in Combination With Azacitidine in Newly Diagnosed Subjects With Acute Myeloid Leukemia Who Are Ineligible for Intensive Chemotherapy in China
Brief Title: Study to Assess Adverse Events and Change in Disease State of Oral Venetoclax in Combination With Subcutaneous (SC) Azacitidine in Newly Diagnosed Adult Participants With Acute Myeloid Leukemia (AML) Who Are Ineligible for Intensive Chemotherapy in China
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M21-569
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia; AML; Venetoclax; Venclexta; Azacitidine; Treatment Naïve AML; Untreated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax in Combination with Azacitidine (Experimental): Participants will receive oral tablet venetoclax dose ramp-up only in Cycle 1 Days 1-3 until target dose is reached. Particpants will then receive oral tablet venetoclax at the target dose every day (QD) on Cycle Days 1 - 28 plus Azacitidine through subcutaneous injection (SC) QD on Cycle Days 1 - 7 (28-day cycle).
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — Tablet: Oral
  Other Names: ABT-199; GDC-0199; Venclexta
Drug: Azacitidine — Subcutaneous Injection (SC)

SUMMARY:
Acute myeloid leukemia (AML) is one of the most aggressive blood cancers, with a very low survival rate and few options for participants who are unable to undergo intensive chemotherapy, the current standard of care. This study is to evaluate how safe the combination of azacitidine and venetoclax is and how effective the combination of azacitidine and venetoclax is in adult participants with acute myeloid leukemia (AML), in China. Adverse events and change in disease state will be assessed.

The combination of azacitidine and venetoclax is being evaluated in the treatment of acute myeloid leukemia (AML). Participants will receive azacitidine with increasing doses of venetoclax. Adult participants with a diagnosis of AML will be enrolled. Around 40 participants will be enrolled in the study in approximately 30 sites in China.

At cycle 1 during ramp-up period, participants will receive venetoclax oral tablets once daily in increasing doses until the study dose is achieved on day 3. Then ventoclax oral tablets will continue once daily thereafter. Azacitidine will be given by subcutaneous injection (SC) for 7 days beginning on Day 1 of each 28-day cycle.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of Acute myeloid leukemia (AML) diagnosis by World Health Organization (WHO) criteria, have a projected life expectancy of at least 12 weeks, previously untreated, and ineligible for treatment with intensive chemotherapy.
* Participant must be considered ineligible for induction therapy defined by the following:

  * >= 75 years of age
  * >=18 to 74 years of age with at least one of the following comorbidities:

    * Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3.
    * Cardiac history of congestive heart failure requiring treatment or ejection fraction <= 50% or chronic stable angina.
    * Diffusing capacity of the lung for carbon monoxide (DLCO) <= 65% or forced expiratory volume during the first second (FEV1) <= 65%.
    * Creatinine clearance >= 30 mL/min to < 45 mL/min.
    * Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × upper limit of normal (ULN).
    * Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy.
* Must meet the laboratory requirements per the protocol.
* Must have an ECOG performance status of:

  * 0 to 2 for subject ≥ 75 year of age; or
  * 0 to 3 for subject ≥ 18 to 74 years of age.
* Female participant must not be pregnant or breastfeeding and is not considering becoming pregnant or donating eggs during the study or for approximately six months after the last dose of study drug.
* Female participants of childbearing potential must agree to use at least 1 protocol-specified method of birth control and male participants, if sexually active with female partner(s) of childbearing potential, must agree to practice the protocol-specified contraception.

Exclusion Criteria:

* History of any malignancies within 2 years prior to study entry with exception noted in the protocol.
* Have received any investigational drug 30 days prior to the first dose of study drug.
* Have received strong and/or moderate CYP3A inducers within 7 days prior to initiation of study treatment.
* Must not have received treatment with the following:

  * An hypomethylating agent (HMA), venetoclax, and/or any chemotherapeutic agent for myelodysplastic syndrome (MDS).
  * Prior therapy or experimental therapies for MDS or Acute myeloid leukemia (AML).
* Current participation in another research or observational study.
* Myeloproliferative neoplasm including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia with or without BCR-ABL1 translocation, and AML with BCR-ABL1 translocation.
* Participant has acute promyelocytic leukemia.
* Participant has known active central nervous system (CNS) involvement with AML.
* Participant has a history of malabsorption syndrome or other condition that precludes enteral route of administration.
* Participant has known HIV infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax). HIV testing will be performed at Screening, only if required per local guidelines or institutional standards.
* Active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) with high viral titers. Participants with HBV inactive carrier status and/or HCV with low viral titers on antivirals (non-exclusionary medications) are eligible.
* Participant has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
* Participant has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition or known hypersensitivity to any of the study medications including excipients of azacitidine that in the opinion of the investigator would adversely affect his/her participating in this study.
* Participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to Approximately 19 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. Treatment-emergent events (TEAEs) are defined as any event that began or worsened in severity after the first dose of study drug. The investigator assesses the relationship of each event to the use of study.
Number of Laboratory Abnormalities from Clinical Laboratory Values (Hematology and Chemistry) | Up to Approximately 19 Months
  Number of Laboratory abnormalities from clinical laboratory values (hematology and chemistry).

SECONDARY OUTCOMES:
Percentage of Participants with Composite Complete Remission (CR [Complete Remission] + CRi [Complete Remission with Incomplete Blood Count Recovery]) Based on the Modified International Working Group (IWG) Criteria for Acute Myeloid Leukemia (AML) | Up to Approximately 19 Months
  CR + CRi is defined as achieving a CR or CRi at any time point during the study prior to the start of post-treatment anti-AML therapies per the modified IWG criteria for AML. CR is defined as absolute neutrophil count (ANC) > 10^3/μL, platelets > 10^5/μL, red cell transfusion independence, and bone marrow with < 5% blasts. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease. CRi is defined as all of the criteria for CR except for residual neutropenia <= 10^3/μL (1000/μL) or thrombocytopenia <= 10^5/μL (100,000/μL). Red blood cell (RBC) transfusion dependence is also defined as CRi.
Percentage of Participants with CR based on the modified IWG criteria for AML | Up to Approximately 19 Months
  CR is defined as absolute neutrophil count (ANC) > 10^3/μL, platelets > 10^5/μL, red cell transfusion independence, and bone marrow with < 5% blasts. Absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- China (18):
  - Peking Union Medical College Hospital (East) - Dongdan Campus /ID# 233179, Beijing, Beijing Municipality
  - Peking University International Hospital /ID# 232254, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center /ID# 231793, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University /ID# 231792, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital /ID# 232059, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 231938, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital /ID# 231444, Shenzhen, Guangdong
  - People's Hospital of Henan Province /ID# 232568, Zhengzhou, Henan
  - Henan Cancer Hospital /ID# 231940, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 233178, Wuhan, Hubei
  - Xiangyang Central Hospital /ID# 232452, Xiangyang, Hubei
  - The First Affiliated Hospital of Soochow University /ID# 232418, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 231442, Nanchang, Jiangxi
  - Qinghai University Affiliated Hospital /ID# 232419, Xining, Qinghai
  - The Second People's Hospital of Yibin /ID# 233180, Yibin, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 232253, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 233704, Wenzhou, Zhejiang
  - Duplicate_The Affiliated Hospital of Guizhou Medical University /ID# 232465, Guiyang

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/